CLINICAL TRIAL: NCT02632045
Title: A randoMized phAse II trIal of fulvestraNt wiTh or Without Ribociclib After Progression on AntI-estrogeN Therapy Plus Cyclin-dependent Kinase 4/6 Inhibition in Patients With Unresectable or Metastatic Hormone Receptor +, HER2 - Breast Cancer (MAINTAIN Trial)
Brief Title: Study of Efficacy of Ribociclib After Progression on CDK4/6 Inhibition in Patients With HR+ HER2- Advanced Breast Cancer
Acronym: MAINTAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melissa K Accordino (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Melissa K Accordino, Assistant Professor of Medicine, Division of Hematology/Oncology, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAP9506
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Breast Cancer; Breast Carcinoma
Keywords: Breast Neoplasms; Breast Cancer; Breast Carcinoma; Breast tumors; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ribociclib (LEE-011)/Fulvestrant (Experimental): LEE-011 is administered orally, 600mg, daily for 3 weeks and 1 week off. Fulvestrant is administered intramuscularly, 500mg, every 2 weeks x 3, then every 4 weeks.
  Interventions: Drug: LEE-011; Drug: Fulvestrant
- Placebo/Fulvestrant (Placebo Comparator): Placebo is administered orally, 600mg daily for 3 weeks and 1 week off. Fulvestrant is administered intramuscularly, 500mg, every 2 weeks x 3, then every 4 weeks.
  Interventions: Drug: Fulvestrant; Drug: Placebo

INTERVENTIONS:
Drug: LEE-011 — 600 mg capsule (3x 200 mg capsules)
  Other Names: ribociclib
  Arms: Ribociclib (LEE-011)/Fulvestrant
Drug: Fulvestrant — 500 mg injection
  Other Names: Faslodex
Drug: Placebo — 600 mg capsule (3x 200 mg capsules)
  Other Names: No other name
  Arms: Placebo/Fulvestrant

SUMMARY:
This is a randomized trial for patients with metastatic hormone receptor (HR)-positive human epidermal growth factor receptor 2 (HER2)-negative breast cancer who have progressed on an aromatase inhibitor plus a CDK4/6 inhibitor (either palbociclib or ribociclib) to either fulvestrant alone or fulvestrant with ribociclib (LEE-011). The purpose of the trial is to determine whether there is continued benefit for patients to remain on a CDK4/6 inhibitor at the time of switching anti-estrogen therapy. As ribociclib and palbociclib have a similar toxicity and drug profile and mechanism of action, the investigators feel that it is appropriate for patients to receive either drug with an aromatase inhibitor prior to randomization.

DETAILED DESCRIPTION:
Despite advances in early detection and therapeutic options, unresectable or metastatic breast cancer remains incurable and is one of the leading causes of cancer-related mortality. Breast cancer is a molecularly heterogeneous disease. This study will be evaluating estrogen receptor (ER) expression positivity and/or progesterone receptor (PgR) positivity of breast cancer with the absence of over-expression or amplification of HER2.

Inhibitors of the cyclin dependent kinases 4 and 6 (CDK4/6) have been developed and demonstrated impressive activity in patients with ER-positive HER2-negative breast cancer with marked improvements in progression free survival. This question is asking whether CDK 4/6 inhibition should be continued with hormone therapy in patients who will be switching their hormone therapy in the metastatic breast cancer setting.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women at least 18 years of age with histologically or cytologically confirmed adenocarcinoma of the breast with unresectable or metastatic disease.
2. Most recent tumor biopsy or surgical resection specimen must be either estrogen-receptor (ER) positive, progesterone receptors (PgR) positive, or both, as defined by immunohistochemistry (IHC) ≥1% (as per the American Society of Clinical Oncology (ASCO)-College of American Pathologists (CAP) guidelines).
3. HER2-negative breast cancer defined as a negative in situ hybridization test or an immunohistochemistry (IHC) status of 0, 1+ or 2+. If IHC is 2+ (i.e. indeterminate), a negative in situ hybridization (Fluorescent in situ hybridization (FISH), Chromogenic in situ hybridization (CISH), or Silver-enhanced in situ hybridization (SISH)) test is required by local laboratory testing. (as per the ASCO-CAP guidelines).
4. Postmenopausal status or receiving ovarian ablation with a GnRH agonist such as goserelin. Postmenopausal status ( is defined by any one of the following criteria:

   * Prior bilateral oophorectomy.
   * Age ≥60 years.
   * Age <60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifen, or ovarian suppression) and follicle stimulating hormone (FSH), luteinizing hormone (LH), and estradiol in the postmenopausal range per local normal If the patient does not meet criteria for postmenopausal status but is receiving ovarian ablation therapy with a gonadotropin-releasing hormone (GnRH) agonist such as goserelin, the patient is eligible for this study, provided that the GnRH agonist is started at least 2 weeks prior to C1D1 of anti-estrogen therapy.
5. Have evidence of measurable or unmeasurable disease.
6. Eastern Cooperative Group (ECOG) performance status of 0 or 1.
7. No prior cdk 4/6 inhibitor (Closed to Accrual). If patient has not previously received letrozole, letrozole will be supplied by Novartis. If previously progressed on letrozole, another aromatase inhibitor that the patient has not previously received is allowed, per standard of care (anastrazole or exemestane, not supplied by study). Ribociclib will be supplied by Novartis. If patient has previously received letrozole, anastrazole, and exemestane, (s)he is not eligible. For scenario 1, patients are allowed to have started the aromatase inhibitor within 4 consecutive weeks prior to protocol registration. For instance, it is acceptable for patient who will be treated with letrozole in scenario #1, to have started letrozole within 4 consecutive weeks prior to protocol registration. No prior fulvestrant allowed.
8. Scenario 2: the patient must have received an aromatase inhibitor (letrozole, arimidex, exemestane) or tamoxifen or fulvestrant plus palbociclib as standard of care or received a CDK4/6 inhibitor (palbociclib or ribociclib or abemaciclib), and demonstrated evidence of disease progression. If the patient was enrolled in a randomized clinical trial involving ribociclib or abemaciclib or palbociclib (such as the MONALEESA or PALOMA series of trials), then it must be known after study discontinuation and unblinding that the patient received the investigational drug and not placebo. Ribociclib or abemaciclib or palbociclib can also be given as standard of care. Documentation of progression and duration of response on aromatase inhibitor or tamoxifen plus CDK 4/6 inhibitor should be provided whenever possible. If patient received prior fulvestrant, exemestane must be the hormone therapy backbone in the randomization. If patient received prior exemestane, fulvestrant must be the hormone therapy backbone in the randomization. If neither has been administered, selection of fulvestrant or exemestane in the randomization will be per investigator discretion.
9. Adequate baseline laboratory studies (hematologic and chemistry), including the following parameters:

   * Absolute neutrophil count ≥ 1500 per microliter, Platelets ≥ 75,000 per microliter, Hemoglobin level ≥ 8.0 gm/dL on screening complete blood count.
   * Potassium, sodium, total calcium (corrected only in the case of hypoalbuminemia), magnesium, and phosphorus within normal limits of the local laboratory (screening values can be rechecked after electrolyte repletion and before the first dose of study medication, if necessary).
   * Serum creatinine level ≤ 1.5 mg/dL or estimated glomerular filtration rate > 50 mL/min.
   * In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) should be below 2.5 × the upper limit of normal (ULN). If the patient has liver metastases, ALT and AST should be < 5 × ULN.
   * Total bilirubin ≤ 1.5 x ULN. (In patients with well documented Gilbert's Syndrome, total bilirubin ≤ 3 × ULN with direct bilirubin within normal range.)
   * international normalized ratio (INR) ≤ 1.5
10. a) Written informed consent and HIPAA authorization obtained from the subject/legal representative prior to performing any protocol-related procedures b) Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
11. Must be able to swallow ribociclib and oral aromatase inhibitor, such as letrozole or exemestane.

Exclusion Criteria:

1. Patient has a known hypersensitivity to any of the excipients of ribociclib, aromatase inhibitors (such as letrozole) or fulvestrant
2. Active central nervous system (CNS) disease. History of CNS metastases or cord compression is allowable if the patient has been clinically stable for at least 4 weeks since completion of definitive treatment and is off systemic steroids. In the case of brain metastases, the patient must have stable or improved imaging at least 4 weeks after completion of definitive treatment. If there is evidence of active leptomeningeal disease, the patient is ineligible.
3. Identified as having visceral crisis, lymphangitic spread, or leptomeningeal carcinomatosis. Visceral crisis is not the mere presence of visceral metastases but implies severe organ dysfunction as assessed by symptoms and signs, laboratory studies, and rapid progression of the disease.
4. Received more than 1 prior systemic chemotherapy in the unresectable or metastatic setting. If the patient received 1 prior systemic chemotherapy, the patient is eligible. Having received prior therapies for breast cancer (such as everolimus or experimental agents) does not affect eligibility for this study.
5. Completion of major surgery, chemotherapy, targeted therapy (such as everolimus or experimental agents_ or radiation within 14 days prior to starting investigational drug or has not recovered from major side effects. There is no required washout period from completion of prior anti-estrogen therapy (either scenario) or prior CDK 4/6 inhibitor (if scenario 2) to initiation of ribociclib/placebo and anti-estrogen on trial.
6. Residual acute toxic effects of prior anti-cancer therapy that have not resolved to CTCAE v.4 Grade ≤1. Exception to this criterion: patients with grade 1 taxane-induced neuropathy, any grade of alopecia, amenorrhea or other toxicities not considered a safety risk for the patient as per investigator's discretion, are allowed to enter the study.
7. Presence of a concurrent malignancy or malignancy diagnosed within 5 years of randomization, with the exception of basal or squamous cell carcinoma, non-melanomatous skin cancer, curatively resected cervical cancer, localized prostate cancer treated with curative intent, and stage I colorectal cancer treated with curative resection.
8. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
9. Patient has a known history of HIV infection (testing not mandatory).
10. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality including any of the following:

    * History of myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to study entry
    * Documented cardiomyopathy
    * Patient has a known Left Ventricular Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO).
    * Long QT syndrome or family history of long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

      i. Risk factors for Torsades de Pointe (TdP) including uncorrected hypocalcemia, hypokalemia or hypomagnesaemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia ii. Concomitant medications(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued or replaced by safe alternative medication (e.g. within 5 half-lives or 7 days prior to starting study drug) iii. Inability to determine the QTc interval
    * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade Atrioventricular block (e.g., bifascicular block, Mobitz type II and third degree Atrioventricular (AV) block)
    * Systolic Blood Pressure (SPB) >160 or <90 mmHg.
11. Corrected QT interval (QTcF) > 450 msec (QT interval using Fridericia's correction) on screening electrocardiogram. If QTc prolongation is felt to be related to electrolyte imbalance, an EKG can be repeated after correction of electrolytes. Mean resting heart rate 50-100 bpm (determined from ECG).
12. The presence of any other concurrent severe and/or uncontrolled medical condition that would, in the investigator or treating physician's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol. This includes uncontrolled infections that could potentially be exacerbated by anti-neoplastic treatment, active untreated or uncontrolled fungal bacterial or viral infections, etc.
13. Currently receiving treatment, including medications and herbal preparations, with known strong inducers or inhibitors of cytochrome p450 enzymes CYP3A4/5 medications that have a narrow therapeutic window and are predominately metabolized through CYP3A4/5 or herbal preparations/medications, dietary supplements, which cannot be discontinued prior to receiving investigational drug. Anti-retrovirals, anti-microbials, and anti-arrhythmics are the most common medications that interact with these enzyme. Please refer to Section 5: Pharmaceutical Information and Appendix B for more information and a list of drugs that should not be used concurrently with ribociclib.
14. Patients who are receiving any other investigational agents concurrently or have received investigational agents within 14 days or 5 half-lives of the compound or active metabolites, whichever is longer before the first dose of the study treatment.

15 Patient is concurrently using hormone replacement therapy. 16. Subject is pregnant or nursing. Serum or urine Beta-Human chorionic gonadotropin (HCG) must be checked in all pre- and peri-menopausal patients. (Fulvestrant is pregnancy category D and CDK4/6 inhibitors have demonstrated teratogenicity/fetotoxicity in animal studies.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Accordino, MD, Principal Investigator — Columbia University
Locations (13):
- United States (13):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Northside Hospital, Inc., Atlanta, Georgia
  - Northwestern Medical Hospital, Chicago, Illinois
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Northwell Health/Monter Cancer Center, Lake Success, New York
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Albert Einstein University / Montefiore Medical Center, The Bronx, New York
  - Vanderbilt-Ingham Cancer Center, Nashville, Tennessee
  - University of Wisconsin School of Medicine, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Herbert Irving Comprehensive Cancer Center (HICCC) Clinical Trials Page — https://cancer.columbia.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 169 participants signed a consent form. Of those, 47 were not randomized or did not start due to the following: n=21 were screen failures, n=18 withdrew consent prior to randomization, n=4 were not randomized due to non-progression. n=4 were randomized however withdrew consent prior to treatment initiation and did not start.
Period: Overall Study
Arm/Group | Placebo/Fulvestrant | Ribociclib (LEE-011)/Fulvestrant
Started | 60 | 62
Completed | 59 | 60
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Fulvestrant | Ribociclib (LEE-011)/Fulvestrant | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [51.5 to 65] | 55 [48 to 67] | 57 [50 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 60 | 118
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 14 | 21
  Not Hispanic or Latino | 48 | 46 | 94
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 42 | 46 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 59 | 60 | 119
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Score on a scale] — The ECOG Performance status scale indicates increasing levels of disability. Scores range from 0 (fully active) to 5 death. A higher score indicates a worse outcome.
  A full description of each score: 0 fully active; 1, restricted in strenuous activity; 2, restricted in work activity but ambulatory and capable of self-care; 3, capable of limited self-care; 4, completely disabled; and 5, dead.
  Score on a scale
    ECOG Performance Status Score 0 | 38 | 40 | 78
    ECOG Performance Status Score 1 | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the interval from the time of randomization until objective disease progression (local assessment) or death from any cause. Disease status will be assessed with comprehensive radiographic studies every three treatment cycles (approximately every 12 weeks (+/- 1 week)). Disease progression as assed by RECIST 1.1 defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to approximately 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo/Fulvestrant | Ribociclib (LEE-011)/Fulvestrant
Number analyzed (Participants) | 59 | 60
months | 2.76 [2.66 to 3.25] | 5.29 [3.02 to 8.12]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Evaluation of disease will be made according to RECIST criteria (version 1.1) in patients with measurable disease. As this study will enroll patients with measureable and un-measurable disease as defined by RECIST v1.1, ORR will only be assessed in evaluable patients. ORR = complete response (disappearance of all target lesions; ny pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm) + partial response (At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters).
Time Frame: measured every 12 weeks, up to 6 months
Population: 35 placebo arm and 35 Ribociclib (LEE-011)/Fulvestrant (n=70) analyzed as these 70 participants had measurable disease.
Measure: Number; unit: participants
Arm/Group | Placebo/Fulvestrant | Ribociclib (LEE-011)/Fulvestrant
Number analyzed (Participants) | 35 | 35
participants | 4 | 7

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR defined as the number of participants with complete response (Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm) + partial response (At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters) + stable disease (Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for disease progression, taking as reference the smallest sum of the diameters while on study) at ≥ 24 weeks of follow up per RESIST 1.1 criteria.
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Fulvestrant | Ribociclib (LEE-011)/Fulvestrant
Number analyzed (Participants) | 59 | 60
Participants | 15 | 26

ADVERSE EVENTS:
Time Frame: 30 days following the last dose of treatment, up to 2.5 years
Description: Systematic collection of adverse events at regular investigator assessment.
Arm/Group | Placebo/Fulvestrant | Ribociclib (LEE-011)/Fulvestrant
All-Cause Mortality (participants affected / at risk) | 2/59 | 2/60
Serious Adverse Events (participants affected / at risk) | 0/59 | 4/60
Other Adverse Events (participants affected / at risk) | 59/59 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Fulvestrant (N=59) | Ribociclib (LEE-011)/Fulvestrant (N=60)
Lung Infection (Infections and infestations) | 0 | 2
Skin Infection (Infections and infestations) | 0 | 1
Kidney Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Fulvestrant (N=59) | Ribociclib (LEE-011)/Fulvestrant (N=60)
Anemia (Blood and lymphatic system disorders) | 13 | 14
Neutropenia (Blood and lymphatic system disorders) | 9 | 43
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 15
Alanine aminotransferase increased (Investigations) | 12 | 10
Anorexia (Metabolism and nutrition disorders) | 7 | 6
Aspartate aminotransferase increased (Investigations) | 17 | 15
Constipation (Gastrointestinal disorders) | 5 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 9
QTC Prolongation (Investigations) | 2 | 8
Fatigue (General disorders) | 19 | 20
Headache (Nervous system disorders) | 6 | 5
Hot Flashes (Vascular disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither the complete nor any part of the results of the study carried out under this protocol, nor any of the information provided by the sponsor for the purposes of performing the study, will be published or passed on to any third party without the consent of the sponsor. Any investigator involved with this study is obligated to provide the sponsor with complete test results and all data derived from the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT02632045/Prot_SAP_000.pdf